CLINICAL TRIAL: NCT02516189
Title: Strength Training for Elderlies and Their Effects on Muscle Fatigue and Microcirculation - Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Professor Fernando Figueira Integral Medicine Institute (Other)
Collaborators: Universidade Estadual da Paraiba (Other)
Responsible Party: Principal Investigator, João Guilherme Bezerra Alves, Teaching Director, Professor Fernando Figueira Integral Medicine Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: FEFMM
Record Dates: First submitted 2015-08-03; First posted 2015-08-05 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Aging
Keywords: Microcirculation; Electromyography; Motor Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): group of elderly participants of strength training program
  Interventions: Other: Strength training program
- Group B (No Intervention): group of seniors who did not practice strength training program

INTERVENTIONS:
Other: Strength training program — Strength Training program applied twice a week for sixteen weeks. Each training exercises has a total time of 50 minutes. Warm-up: 5 minutes of stretching. Training: Leg press; Leg Curl; Vertical traction; Chest press; Abdominal crunch; Lower back. Gametherapy.
  Relaxation: 5 minutes of stretching.
  Arms: Group A

SUMMARY:
The purpose of this study is to verify the effects of a strength training program on functional capacity, muscle performance and microcirculation in the elderly.

DETAILED DESCRIPTION:
Purpose

The primary research question is:

Do muscular strength training programs can improve functional capacity, muscle performance and microcirculation in the elderly? Hypothesis: Strength training program will promote electromyographic changes during the development of peripheral muscle fatigue and microcirculatory blood flow contributing to functional autonomy.

Secondary Research Questions

1. Does the strength training program in the elderly improve the standard of electromyographic fatigue? Hypothesis: Elderly practitioners of strength exercise program showed increased neuromuscular efficiency and electromyographic fatigue index.
2. Do the strength training program in the elderly improve peripheral microcirculation? Hypothesis: A regular program of strength exercise in the elderly increases the blood flow in peripheral microcirculation changing the process of muscle fatigue. These biomechanical and physiological changes contribute to increased functional autonomy and reducing the risk of falls in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* sedentary elderly
* individuals who have physical and medical conditions to perform strength training
* individuals who participate in the Open University Maturity Program

Exclusion Criteria:

* individuals who do not have physical and medical conditions to perform strength training

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in elderlies's microcirculatory blood flow after 4 months | 4 months
  The blood flow in the microcirculation in the elderly will be measured by laser-doppler flowmetry. The measures blood flow in the microcirculation will be quantified by the reactive hyperemia Post-occlusion protocol (PORH).
Change in elderlies's muscle fatigue after 4 months | 4 months
  muscle fatigue will be quantified by surface electromyography of the muscles of the lower limbs. The electromyographic fatigue threshold and fatigue index will be calculated by the Root Mean Square (RMS) and Median Frequency variables after 4 months.
Change in elderlies's functional capacity after 4 months | 4 months
  The functional capacity of the elderly will be evaluated by the Berg Balance Scale, the Timed up-and-go Test, and Falls Efficacy Scale International (FES-I) after 4 months

SECONDARY OUTCOMES:
Change in elderlies's strength after 4 months | 4 months
  The lower body strength of the elderly will be measured by 30-s chair test stand after 4 months.
Change in elderlies's functional autonomy after 4 months | 4 months
  The functional autonomy of the elderly will be determined by the general functionality index of the Latin American Development Group to Maturity Protocol after 4 months.

CONTACTS AND LOCATIONS:
Overall Officials: Danilo A Vasconcelos, MS, Principal Investigator — Universidade Estadual da Paraiba; João G Alves, PhD, Principal Investigator — Instituto de Medicina Integral Professor Fernando Figueira